CLINICAL TRIAL: NCT01607801
Title: Effect of Reoperation for Recurrence After Open Surgery for Small Umbilical Hernia With Sutured Mesh or Plastic Surgery. A National Hernia Database Study.
Brief Title: Effect of Reoperation for Recurrence After Open Umbilical Hernia Repair
Acronym: UMBI-REC
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Mette M W Christoffersen, Medical Doctor, Zealand University Hospital
Other Study IDs: UMBI-123
Record Dates: First submitted 2012-05-25; First posted 2012-05-30 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Umbilical Hernia
Keywords: umbilical hernia repair; recurrence; choice of suture; mesh; mesh/non-mesh
MeSH Terms: conditions — Hernia, Umbilical; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- non-absorbable suture NAS: having their umbilical hernia repaired with NAS
- Long-term-absorbable suture (LAS): patients having their umbilical hernia repair with LAS
- Absorbable sutures (AS): patients having their umbilical hernia repair with AS
- Mesh repair: Patients having umbilical hernia mesh repair

SUMMARY:
background Operation for small umbilical hernias is one of the most common surgical procedures, but the best surgical technique, including the choice of suture or mesh remains unknown.

It is well known that using non-absorbable sutures in closure of the abdomen, diminishes the risk of incisional hernias and wound healing problems.It has also been found that the use of resorbable suture in fixation of the mesh in Lichtesteins procedure leads to greater risk of recurrence of the hernia. Furthermore, it has been stated in smaller studies, that the use of the mesh in open operation for a small umbilical hernia has lower risk of recurrence (approx. 1-3%) than sutured repair (10-12 %). However, the scientific literature is deficient, with few patients.

The purpose of this study is to describe reoperation rate of recurrence after small umbilical hernias, depending on choice of sutures in both regular repair and in mesh repair.

Hypothesis: sutured repair with non-absorbable suture has lower recurrence rates than with other types of sutures, whereas mesh repair has even lower recurrence rates in small umbilical hernia repairs.

DETAILED DESCRIPTION:
National prospective registry study with data from the Danish ventral hernia Database (DVHD) and the National Patient Register (LPR) in patients undergoing open to umbilical or epigastric hernia repair during the period 1 January 2007 to 31 December 2010.

Apart from operator-registered perioperative data from DVHD, operations can be characterized with different types of sutures, choice of mesh and other relevant information, with possible impact on long-term outcome after surgery, including recurrence.

There will be used frequency analyzes and Kaplan Meyer statistics, supplemented by multivariate Cox regression analysis, as well as non-parametric statistics.

Eligibility criteria: OPen mesh or sutured repair for small umbilical hernias from 1th of January 2007 to 31th of December 2010.

Outcome measures: Reoperation as a surrogate for recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Mesh or non-mesh umbilical hernia repair hernia defect size max. 2 cm.

Exclusion Criteria:

* bigger defect than 2 cm. laparoscopic repair

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Danish patients undergoing umbilical hernia repair, mesh/non-mesh, under 2 cm. in the study period 1. january 2007 to 31. december 2010.
Sampling Method: Non-Probability Sample
Enrollment: 4847 (Actual)
Dates: Start 2007-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
reoperation as surrogate for recurrence | 4 years
  all patients having hernia recurrence measured as reoperation, cross-checked with National Patient Register

CONTACTS AND LOCATIONS:
Locations (1):
- Koege Sygehus, Koege, Denmark

REFERENCES:
- [Derived] Christoffersen MW, Helgstrand F, Rosenberg J, Kehlet H, Bisgaard T. Lower reoperation rate for recurrence after mesh versus sutured elective repair in small umbilical and epigastric hernias. A nationwide register study. World J Surg. 2013 Nov;37(11):2548-52. doi: 10.1007/s00268-013-2160-0. PMID 23887595